CLINICAL TRIAL: NCT03645213
Title: Comparision of Two Different Distraction Methods on Pain and Fear During Venipuncture in School-Age Children: A Randomized Controlled Trial
Brief Title: Two Different Distraction Methods on Pain and Fear During Venipuncture in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Demet İnangil, PhD, Assistant Professor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10840098-604.01.01-E.40485
Record Dates: First submitted 2018-08-10; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Venipuncture Site Reaction; Procedural Complication; Nursing Caries
Keywords: School-age children; pain; fear; venipuncture; distraction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial study was conducted on 120 school-age children (7 -12 years of age) with pain and fear of venipuncture. The children were randomized according to their arrival in the biochemistry laboratory; the first, second, and third children were assigned VR distraction group with a headset (n=40), non-VR distraction group on a tablet computer screen (n=40) and no distraction group (n=40), respectively. The data collection was carried out using the children identification form, Wong-Baker FACES Pain Rating Scale evaluating the pain and Childrens' Fear Scale evaluating the fear. The outcomes reported by the children, parent, and observer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality (VR) (Experimental): Children were asked which cartoon they wanted to watch and it was prepared. The cartoons began to be shown a minute before venipuncture and lasted about 4 minutes. The procedure and reason were explained to the child before each step of the venipuncture process such as apply a tourniquet, insert and remove the needle. The parent stopped on the left side of the child's. The display was a head-mounted VR box in the VR group.
  Interventions: Device: Virtual Reality Box
- Non- Virtual Reality (VR) (Experimental): Children were asked which cartoon they wanted to watch and it was prepared. The cartoons began to be shown a minute before venipuncture and lasted about 4 minutes. The procedure and reason were explained to the child before each step of the venipuncture process such as apply a tourniquet, insert and remove the needle. The parent stopped on the left side of the child's. The display was a computer tablet in the non-VR group. The computer tablet was the 10 centimeters far from the child.
  Interventions: Device: Tablet Computer
- Control (No Intervention): There was no additional intervention in the control group. Venipuncture procedures was the same other groups. The procedure and reason were explained to the child before each step of the venipuncture process such as apply a tourniquet, insert and remove the needle. The parent stopped on the left side of the child's.

INTERVENTIONS:
Device: Virtual Reality Box — Virtual Reality box, a head-mounted display with stereo earphones transmits the cartoon image onto screens in front of the child's eyes. It was showed on Samsung Galaxy Note5 phone and Samsung Gear VR box /SM-R323N.
  Arms: Virtual Reality (VR)
Device: Tablet Computer — The tablet computer is a device that children watch on a 7-inch screen.
  Arms: Non- Virtual Reality (VR)

SUMMARY:
Objective: Needle-related procedures (venipuncture, vaccine injections) are the most common source of pain and fear, and generally experienced in childhood for the first time. This study was designed to determine the effects of watching cartoon films on non-VR and VR virtual reality on pain and fear during venipuncture in school-age children and to compare these two methods.

Method: This randomized controlled trial study was conducted on 120 school-age children (7 -12 years of age) with pain and fear of venipuncture. The children were randomized according to their arrival in the biochemistry laboratory; the first, second, and third children were assigned VR distraction group with a headset (n=40), non-VR distraction group on a tablet computer screen (n=40) and no distraction group (n=40), respectively. The data collection was carried out using the children identification form, Wong-Baker FACES Pain Rating Scale evaluating the pain and Childrens' Fear Scale evaluating the fear. The outcomes reported by the children, parent, and observer.

DETAILED DESCRIPTION:
Introduction: Needle procedures (eg, venipunctures, vaccine injections) are the most common and generally experienced in childhood for the first time. Children often describe needle procedures as the most painful and fearful intervention in the healthcare. The pain and fear of injections may affect the children psychologically and lead to situations such as refusal of interventions in children. Besides, these effects can disrupt the communication between nurses and children and cause distress to parents. Unmitigated pain during these procedures may increase fear which in turn can exacerbate future pain in an escalating relationship. However, there are no studies on the techniques applied to reduce pain and fear during venipuncture in school-age children, nor are there any comparing watching cartoon films and virtual reality. This study was carried out to determine the effects of watching cartoon films on non-VR and VR virtual reality on pain and fear during venipuncture in school-age children and to compare these two methods.

Study design A randomized controlled clinical trial was conducted.

The following hypotheses (H) were tested in this study:

H1. Watching cartoon films by non-VR distractor to children during venipuncture would be effective in controlling pain and fear.

H2. Watching cartoon films by VR distractor to children during venipuncture would be effective in controlling pain and fear.

Sample and Setting This study was conducted with 120 children, studying at the at the Biochemical Laboratory of Medipol University Hospital, Turkey between September 2017-April 2018. The sample included in the study were required to meet the eligibility criteria of being between 7-12 years old, a physician order was placed for blood sample, no current acute pain, no cognitive or severe physical disability, no communication difficult, blood sample was taken in the first attempt and consent of the parents for the child to take part in the research. The sample consisted of 120 out of the 147 children aged. Among the 27 children not included the sample group.

Childrens were divided into 3 groups. The children were randomized according to their arrival in the biochemistry laboratory; the first, second, and third children were assigned VR group (n=40), non-VR group (n=40) and control group (n=40), respectively. The outcome measures were the level of pain and fear by the children, the parent and blinded research observer, immediately after venipuncture procedures.

Data Collection Form Data collection was carried out using (a) the Children Identification Form prepared by the authors, (b) Wong-Baker FACES Pain Rating Scale and (c) Childrens' Fear Scale.

Procedure The procedure and reason were explained to the child before each step of the venipuncture process such as apply a tourniquet, insert and remove the needle. The parent stopped on the left side of the child's in all groups. The display was a head-mounted VR box in the VR group. The computer tablet was the 10 centimeters far from the child in the non-VR group.

ELIGIBILITY:
Inclusion Criteria:

* being between 7-12 years old,
* a physician order was placed for blood sample,
* no current acute pain,
* no cognitive or severe physical disability,
* no communication difficult,

Exclusion Criteria:

* the blood sample cannot be taken in the first attempt
* no consent of the parents for the child to take part in the research

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Measure | Immediately after venipuncture
  Used for the pain intensity during the procedure was the Wong-Baker FACES Pain Rating Scale (WB-FBRS) which is represented by six animated faces arranged side by side from the worst pain to the mildest one (0-5). The range of painfulness from the smiling "no pain" (0 points) to the crying face of "the worst pain" (5 points) translated into the Turkish language

SECONDARY OUTCOMES:
Fear Measure | Immediately after venipuncture
  The Childrens Fear Scale (CFS) is used to measure the anxiety or fear level of the children. The CFS is developed by McMurtry et al. 2011 based on the Faces Anxiety Scale to measure anxiety or fear in adults in the intensive care unit. The scale faces were drawn by a graphic artist according to the facial muscle changes involved in a fearful expression. The one-item scale consists of a row of five sex neutral faces ranging from a no fear (neutral) face on the far left to a face showing extreme fear on the far right.

CONTACTS AND LOCATIONS:
Overall Officials: Merdiye Şendir, Proffessor, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mutlu B, Balci S. Effects of balloon inflation and cough trick methods on easing pain in children during the drawing of venous blood samples: a randomized controlled trial. J Spec Pediatr Nurs. 2015 Jul;20(3):178-86. doi: 10.1111/jspn.12112. Epub 2015 Mar 28. PMID 25817062
- [Result] Karakaya A, Gozen D. The Effect of Distraction on Pain Level Felt by School-age Children During Venipuncture Procedure--Randomized Controlled Trial. Pain Manag Nurs. 2016 Feb;17(1):47-53. doi: 10.1016/j.pmn.2015.08.005. Epub 2015 Oct 12. PMID 26459008